CLINICAL TRIAL: NCT05117944
Title: The Effect of Drama-supported "Patient Role" Experience on Nursing Students' Empathy and Altruism Levels: a Randomized Controlled Study
Brief Title: Drama-supported Patient Role Experience of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulden Basit (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Sponsor-Investigator, Gulden Basit, Necmettin Erbakan University Faculty of Nursing, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21129001
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Nursing Students; Empathy; Altruism; Patient
Keywords: nursing; nursing student; nursing education; empathy; altruism; patient; drama
MeSH Terms: conditions — Altruism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drama (Experimental): Students in the intervention group will act as the patient and act out the case given to them. Nursing care to be provided by a professional nurse to the student who will play the role of the patient in line with the case content includes helping the patient (student) eat, perform personal hygiene (oral care, etc.), dress and move. The case content will not be shared with the students in advance, and the student will not need to make any preliminary preparations. However, ten minutes before the start of the practice, the situations that are expected to be portrayed as the patient specified in the case will be explained to the students. The skills laboratory will be used as three separate patient rooms (with two or three patients), in which students in the role of inpatient will receive care from a professional nurse. Each student will experience the patient role only once.
  Interventions: Other: drama-supported "patient role" experience
- Control (No Intervention): Students in the control group will fill in the datasheet, Altruism Scale and Empathy Scale simultaneously with the intervention group, without any intervention, and then the Altruism Scale and Empathy Scale at the 1st and 3rd months.

INTERVENTIONS:
Other: drama-supported "patient role" experience — The students participated in 3 hours of drama activities and played the role of a patient whose basic needs such as nutrition, dressing and oral care were met by the nurse, lying down for 4 hours in the skills laboratory.
  Arms: Drama

SUMMARY:
"Empathy", one of the skills required by the nursing profession, has an important place in the patient-nurse relationship. Considered as the most basic motivation of altruistic behaviour, empathy requires recognizing the emotional states of others and understanding their needs. The aim of this study is to determine the effect of drama-supported "patient role" experience on nursing students' empathy and altruism levels. Method: This research was designed as a pretest-posttest regular parallel-group, randomized controlled experiments. The research will be carried out with students studying in Necmettin Erbakan University Faculty of Nursing, 2nd grade, without a history of hospitalization and chronic disease and who agreed to participate in the research. Data will be collected using the Datasheet, Altruism Scale, and Jefferson Empathy Scale for Nursing Students (JESNS). The data will be analyzed in the SPSS program.

DETAILED DESCRIPTION:
This research was designed as a pretest-posttest regular parallel-group, a randomized controlled experimental study to determine the effect of drama-supported "patient role" experience on nursing students' empathy and altruism levels.

The hypotheses of the research; H1_0: The nursing students' empathy levels who experienced the drama-supported "patient role" were not different from those in the control group.

H1_1: The nursing students' empathy levels who experienced the drama-supported "patient role" were different from those in the control group.

H2_0: The altruism levels of the nursing students who experienced the drama-supported "patient role" were not different from those in the control group.

H2_1: The altruism levels of the nursing students who experienced the drama-supported "patient role" differed from those in the control group.

The place and features of the research:

The research will be carried out at Necmettin Erbakan University Faculty of Nursing. There is a nursing practice skill laboratory consisting of 3 rooms and ten beds in the faculty building. Accordingly, it is appropriate to research a laboratory environment.

Study group:

The study group consists of second-year students (N=158) studying at Necmettin Erbakan University, Faculty of Nursing, Department of Nursing in the 2021-2022 academic year.

The ethical dimension of research Necessary permissions were obtained from Necmettin Erbakan University Meram Medical Faculty, Non-Pharmaceutical and Medical Device Research Ethics Committee (date/decision no: 22.05.2020/2536) and Necmettin Erbakan University Nursing Faculty for the implementation of the study. Written permission was obtained from Aygül Yanık, who conducted the Jefferson Empathy Scale for Nursing Students (2014). Written permission was obtained from Mr Ümmet, Ekşi, and Otrar, who developed the Altruism Scale (2013). Informed Consent will be obtained from the students participating in the research before starting the application. After the implementation of the study, training on empathy and altruism in nursing will be organized, and a certificate of participation will be given to all students participating in the research.

Data collection:

The data of the research will be collected between November 2021 and February 2022. Students who accept the study will fill out the datasheet, Altruism Scale (pretest) and Jefferson Empathy Scale for Nursing Students (pretest) in the classroom environment. Students will be randomly assigned to the intervention and control groups, stratified by gender (random.org will generate random numbers). Students in the intervention group will attend 3-hour drama workshops before the "patient role" experience. After the students experience the patient role under the supervision of researchers in the skills laboratories of Necmettin Erbakan University Nursing Faculty, they will refill the Altruism Scale and the empathy scale as a posttest (1 month after the intervention). The scales will be filled again at the end of the 3rd month to monitor the change in the empathy and altruism levels of the students. Students in the control group will fill out the Introductory Characteristics Form, the Altruism Scale and the Empathy Scale simultaneously with the intervention group, without any intervention, and then the Altruism Scale and the Empathy Scale at the end of the 1st and 3rd months. Due to ethical reasons, after the research data is collected, willing students in the control group will experience the patient role.

Statistical analysis of data:

Parametric or nonparametric tests will be applied according to descriptive statistics such as the number per cent mean standard deviation in the SPSS (Statistical Package For Social Science) program and normality test results of the data. The results obtained will be interpreted according to the significance level of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* second-year nursing student

Exclusion Criteria:

* have a history of hospitalization
* have a chronic disease
* working as a nurse

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
The Jefferson Empathy Scale for Nursing Students | Change from empathy levels of students at one and third months from baseline
  1. The Jefferson Empathy Scale for Nursing Students: Hojat et al. (2001) for physicians and adapted for nursing students by Ward (2009). The scale for nursing students was adapted to Turkish by Yanık and Saygılı (2014), and its validity and reliability were established. The original scale consisted of 20 items and three sub-dimensions. The Turkish version consists of 3 sub-dimensions (catching the patient's point of view, compassionate care, putting yourself in the patient's place) and 18 items, as in the original. The scale is a 7-point Likert type (1=strongly disagree, 7=strongly agree) and is scored between 18-126. Items 1, 3, 6, 7, 8, 11, 12, 14, 18 and 19 are reverse scored on the scale. The higher the score, the higher the level of empathy. It has been reported that the total Cronbach alpha value of the scale was calculated as 0.73. This scale will be filled in during the pre-test, post-test and follow-up phases of the research
Altruism Scale | Change from alturism levels of students at one and third months from baseline.
  2. Altruism Scale: The scale developed by Ümmet, Ekşi, and Otrar (2013) to measure the altruistic behaviours of individuals has seven sub-dimensions (participation in voluntary activities, financial assistance, assistance in traumatic situations, assistance to the elderly/patients, assistance based on physical strength, in education process). It is a 5-point Likert-type scale (1=I strongly disagree, 2=Disagree, 3=I am undecided, 4=I agree, 5=I totally agree) consisting of 38 items (help, help arising from a sense of closeness) and 38 items. The total Cronbach Alpha value of the scale was stated as 0.81. There is no reverse item and cut-off point in the scale, and a high score (min: 38- max: 190) indicates high altruism. This scale will be filled in during the pre-test, post-test and follow-up stages of the research.

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Basit, RN, PhD, Principal Investigator — Necmettin Erbakan University Faculty of Nursing
Locations (1):
- Necmettin Erbakan University Faculty of Nursing, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No